CLINICAL TRIAL: NCT05875207
Title: Physical Therapy Integrated With Mindfulness for Patients With Chronic Musculoskeletal Pain and Long-Term Opioid Treatment
Brief Title: Physical Therapy Integrated With Mindfulness for Patients With Chronic Pain and Opioid Treatment
Acronym: PT-IN-MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Florida (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jake Magel, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 159762; 1R01AT012229-01 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-05-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Pain, Musculoskeletal; Opioid Use; Physical Therapy
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: This is a multi-site feasibility randomized clinical trial.
Who Masked: Investigator
Masking Description: Lead statistician is also masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Evidence based physical therapy combined with mindfulness (Low-Intensity) (Experimental): Physical therapists randomized to this arm will receive a manual on how to integrate MORE; mindfulness, mindful reappraisal, and mindful savoring savoring into routine outpatient physical therapy for patients with chronic musculoskeletal pain and long-term opioid treatment.
  After 4 weeks to review the manual, the physical therapist's competency will be assessed during mock patient encounters using trained actors as standardized patients.
  Patients with chronic musculoskeletal pain and long-term opioid treatment who seek care from a physical therapist in this arm will be approached to participate in the study. If eligible and willing to participate in the study they will be asked questions about pain and opioid use before, and after treatment. We plan on enrolling 2 patients for each physical therapist.
  Interventions: Behavioral: Mindfulness based practice
- Standard physical therapy (Other): Physical therapists randomized to this arm will deliver routine treatment for someone with chronic musculoskeletal pain and long-term opioid treatment.
  Patients with chronic musculoskeletal pain and long-term opioid treatment who seek care from a physical therapist in this arm will be approached to participate in the study. If eligible and willing to participate in the study they will be asked questions about pain and opioid use before, during and after treatment. We plan on enrolling 2 patients for each physical therapist.
  Interventions: Behavioral: Control/Standard Physical Therapy
- Evidence based physical therapy combined with mindfulness (High-Intensity) (Experimental): Physical therapists randomized to this arm will receive 13 hours of training. The first 6 hours consists of prerecorded didactic lectures that the physical therapist can view on their own time. After viewing the lectures, participants will attend 6.25 hours of live experiential instruction to promote trainee competence in providing mindfulness, mindful reappraisal, and mindful savoring after which the participating physical therapist's competency will be assessed during mock patient encounters using trained actors as standardized patients. .
  Patients with chronic musculoskeletal pain and long-term opioid treatment who seek care from a physical therapist in this arm will be approached to participate in the study. If eligible and willing to participate in the study they will be asked questions about pain and opioid use before, and after treatment. We plan on enrolling 2 patients for each physical therapist.
  Interventions: Behavioral: Mindfulness based practice

INTERVENTIONS:
Behavioral: Mindfulness based practice — Physical therapists who are randomized to this arm will receive mindfulness training. This training will teach physical therapists to use the following with their patients: 1) use mindfulness to strengthen self-regulation of habitual and compulsive opioid use, and to mitigate pain by reinterpreting these experiences as innocuous sensory information, 2) use reappraisal to reframe stressors and maladaptive thoughts to decrease negative emotions and engender meaning in life, 3) use savoring of pleasant events and pleasurable sensations to enhance positive emotions and reward and, 4) to integrate mindfulness, reappraisal and savoring with evidence-based physical therapy.
  Arms: Evidence based physical therapy combined with mindfulness (High-Intensity); Evidence based physical therapy combined with mindfulness (Low-Intensity)
Behavioral: Control/Standard Physical Therapy — Physical therapists randomized to this arm will receive no additional training and will provide standard care to patients with chronic musculoskeletal pain and long-term opioid treatment. Patients with chronic musculoskeletal pain and long-term opioid treatment who seek care from a physical therapist in this arm will be approached to participate in the study. If eligible and willing to participate in the study they will be asked questions about their pain and opioid use before and after treatment. We plan on enrolling 2 patients for each physical therapist.
  Arms: Standard physical therapy

SUMMARY:
This study will use multiple methods to assess the feasibility of conducting a fully powered multisite clinical trial to test the effectiveness of integrating mindfulness-based interventions into physical therapy for patients with chronic musculoskeletal pain and long-term opioid treatment.

First, researchers will develop a manual for training physical therapists to provide mindfulness-based interventions to patients with chronic musculoskeletal pain and long-term opioid treatment. Next, the researchers will evaluate the competency of physical therapists to provided mindfulness-based interventions after being randomized to one of 3 different mindfulness training arms. Patients scheduled for physical therapy with the randomized physical therapists will be invited to enroll in the study. These patients will be asked to complete a variety of patient reported outcomes including self-reported average pain and the the amount of prescription opioid pain medication taken.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain is a leading cause of years lived with disability world-wide and the costliest health condition in the United States. An estimated 20%-30% of persons with chronic musculoskeletal pain use opioids for pain management. In recent years, the prevalence of long-term opioid treatment (LTOT) has increased in patients with musculoskeletal pain. Physical therapy (PT) is a common nonpharmacologic treatment recommended for chronic musculoskeletal pain. Studies suggest PT for musculoskeletal pain may reduce the likelihood of initiating opioid therapy and may protect against LTOT, but the role of PT as part of a multi-modal strategy to manage patients with chronic musculoskeletal pain and LTOT has not been investigated. Combining exercise-based interventions with mindfulness practices is effective for patients with chronic musculoskeletal pain, and engaging in mindfulness practices leads to a reduction in opioid dose in patients with chronic pain and LTOT. This is a feasibility study that will assess effectiveness of physical therapists in managing patients with chronic musculoskeletal pain and LTOT using mindfulness practices. the results of an aim may result in changes to the procedures of a subsequent aim.

This study is organized into three Aims that will be conducted consecutively.

Aim #1: is to refine and manualize physical therapist-led mindfulness-based interventions integrated with evidence-based PT (I-EPT) for patients with chronic musculoskeletal pain and LTOT. Our approach will use semi-structured interviews of 15 patients and 15 physical therapists to refine I-EPT.

Aim #2: Evaluate different intensities of a physical therapist training programs for the refined I-EPT treatment protocol. Our approach will be to randomize 45 physical therapists to 1 of 3 training arms (no training; low-intensity training; high-intensity training).

Aim #3: Evaluate the feasibility of the I-EPT intervention across domains of the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework. We anticipate 90 patient participants will be enrolled onto the schedules of the randomized physical therapists in Aim 2. Semi-structured qualitative interviews will be conducted. For these interviews there will be separate cohorts of 27 participants from Utah and 27 from Florida. Each cohort will contain approximately 8 physical therapists (4 each from the HIghIT and LowIT programs), 13 patients and 7 between support staff, and clinic managers.

ELIGIBILITY:
Aim 1

Physical Therapist Inclusion Criteria:

* Employed at least .50 FTE (Full Time Equivalent)
* Self Report managing patients with chronic musculoskeletal conditions

Exclusion Criteria: None

Aim 2 and 3

Physical Therapist Inclusion Criteria:

* Employed at least .50 FTE (Full Time Equivalent)
* Self Report managing patients with chronic musculoskeletal conditions

Physical Therapist Exclusion Criteria:

* -Attended any experiential (i.e., practice sessions with real or simulated patients) mindfulness training to be used for patient care
* Attended any patient care specific mindfulness training lasting more than 3 hours.
* Self-report using mindfulness interventions such as savoring and cognitive reappraisal (core components of MORE) as a primary intervention strategy for the majority of their caseload for patients with chronic musculoskeletal conditions.

Aims 1, 2 and 3

Patient Inclusion Criteria:

* Age 18-75
* English Speaking
* Diagnosis of musculoskeletal pain condition involving the spine and/or peripheral joint(s)
* Current musculoskeletal pain present for greater than or equal to 3 months.
* Use of prescription opioids for most of the last 90 days (self-report)

Patient Exclusion Criteria:

* Currently pregnant
* Currently receiving mind-body treatment for musculoskeletal pain from a healthcare provider (e.g. PT, chiropractic, massage therapy, etc)
* Currently receiving treatment for substance use disorder
* Musculoskeletal pain condition related to a fracture or surgical procedure in the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Aim #2: Mindfulness Oriented Recovery Enhancement fidelity measure | 6 - 8 weeks after I-EPT live training
  Mindfulness Oriented Recovery Enhancement fidelity (Modified MORE-FM) Version 2.0 measure score during post-training competency assessment of physical therapists (physical therapists randomized to High and Low Intensity training groups)
  9 item scale - each item scored 0-6. Scores are summed and averaged.
Aim #3: Opioid MMEs on Timeline followback (TLFB) | 12 weeks
  Percentage of TLFBs collected at 12 weeks
  The TLFB collects number of morphine milligram equivalents taken by the patient over the past 4 weeks
Aim 3: PEG (Pain, Enjoyment, General activity) | 12 weeks
  Percentage of The Pain, Enjoyment and General Active (PEG) scales collected at 12 weeks
  The PEG measures pain intensity, enjoyment of life and general activity each on a 0 - 10 with higher scores indicating worse pain impact. The score is the average of all items.

SECONDARY OUTCOMES:
Aim #1 Qualitative Interviews | 1 month
  Semi-structured qualitative interviews will be conducted with patients and physical therapists after they review a mindfulness treatment protocol. Analysis will generate qualitative themes that will be used to modify the treatment protocol in preparation for Aim #2.
Aim #2: Physical therapist retention (competency assessment) | 6 - 8 weeks after I-EPT live training
  Percent of physical therapists who attend the competency assessment.
Aim #2: Randomized physical therapists | At recruitment
  Percentage of physical therapists invited who consent to be randomized
Aim #2: Physical therapist enrollment | At recruitment
  Percent of physical therapists presented the study who choose to enroll in the study
Aim #3: Opioid MMEs on Timeline followback (TLFB) | Baseline 6 and 12 weeks
  The TLFB collects number of morphine milligram equivalents taken by the patient over the past 4 weeks
  We will calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
Aim 3: PEG (Pain, Enjoyment, General activity) | baseline, 6 and 12 weeks
  The PEG measures pain intensity, enjoyment of life and general activity each on a 0 - 10 with higher scores indicating worse pain impact. The score is the average of all items.
  We will calculate the change from baseline to 6 and from baseline to 12 weeks
Aim #3 Patient Reported: Pain Catastrophizing Scale (PCS) short form | baseline, 6 and 12 weeks
  Percentage of PCS short form scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  Scores range 0- 24. Higher scores mean greater catastrophizing.
Aim #3 Patient Reported: Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 6b (PROMIS-6b) | baseline, 6 and 12 weeks
  Percentage of PROMIS-6Bs collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  PROMIS-6b is reported as a T-Score with a mean of 50 and a SD of 10
Aim #3 Patient Reported:Patient Reported Outcomes Measurement Information System (PROMIS)PROMIS Sleep Disturbance Short Form 6a | baseline, 6 and 12 weeks
  Percentage of PROMIS Sleep Disturbance Short Form 6As collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  Reported as a T-Score with a mean = 50 and a SD = 10
Aim #3 Patient Reported: Patient Health Questionnaire-2 (PHQ-2) | baseline, 6 and 12 weeks
  Percentage of PHQ-2 scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  Scores range from 0-6. Higher scores mean greater likelihood of depression
Aim #3 Patient Reported: Generalized Anxiety Disorder-2 (GAD-2) | baseline, 6 and 12 weeks
  Percentage of GAD-2s collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  2 items summed range 0 - 6. Higher score mean greater likelihood of anxiety
Aim #3 Patient Reported: Patient Global Impression Scale-Change | 6 and 12 weeks
  Percentage of Patient Global Impression Scale-Change scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  Scores range from 0 - 7 with higher score equating to greater improvement in condition
Aim #3 Patient Reported: Pain Self-Efficacy Questionnaire (PSEQ) | baseline, 6 and 12 weeks
  Feasibility: Percentage of PSEQ scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  PSEQ scores range from0 - 60 with higher scores indicating greater levels of confidence in dealing with pain
Aim #3 Patient Reported: Mindfulness-Five Facet Mindfulness Questionnaire (FFMQ) | baseline, 6 and 12 weeks
  Feasibility: Percentage of FFMQ scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  FFMQ has15 items and scores range from 15 - 75 higher scores indicate greater mindfulness
Aim #3 Patient Reported: Positive Reappraisal Subscale of Cognitive Emotion Regulation Questionnaire (reappraisal subscale) | baseline, 6 and 12 weeks
  Feasibility: Percentage of reappraisal subscale scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  4 items each scored 1 - 5. Higher the score the more positive reappraisal.
Aim #3 Patient Reported: Savoring Beliefs Inventory | baseline, 6 and 12 weeks
  Percentage of Savoring Beliefs Inventory scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  24 items - Composite scores are obtained by averaging the subscales after rescoring the negatively worded items. Higher scores equate to greater savoring.
Aim #3 Patient Reported: Participant-report health care utilization measures | 4, 8 and 12 weeks
  Measure health care use (imaging,, tests, physician visits, medications)
Aim #3 Patient Reported: Short Assessment of Patient Satisfaction | 6 and 12 weeks
  Percentage of Short Assessment of Patient Satisfaction scores collected at 6 and 12 weeks.
  We will also calculate the scores at 6 and 12 weeks
  7 items. Each item scored 0 - 4 . Reverse score items 1, 3, 5 and 7. Sum scores. Range from 0 (extremely dissatisfied to 7 (extremely satisfied)
Aim #3 Reach: Patients offered and enrolled | At recruitment
  The percentage of patients with chronic muscle condition and long-term opioid treatment offered participation who choose to enroll.
Aim #3 Patient Reported: The International Pain Activity Questionnaire (IPAQ) short form measures physical activity | Baseline, 6 and 12 weeks
  Percentage of IPAQ scores collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
  7 items. Measures metabolic equivalents (METS). Higher score in METS equates to greater activity.
Aim #3. Patient Reported: Working Alliance Inventory - Short Short Revised (WAI-SR) Client Version | 4, 8 and 12 weeks
  Percentage of WAI-SR scores collected at 4, 8 and 12 weeks
  We will also calculate the change from 4 to 8 weeks and the change from 4 to 12 weeks.
  12 items. Higher scores indicate better therapeutic alliance.
Aim #3 Reach: Physical therapists with enrolled patients | At recruitment
  The percentage of physical therapists who have a patient enrolled on their schedule
Aim #3 Effectiveness: REDCap Outcomes Collected | 12 weeks
  The percentage of all patient reported outcome measures collected using REDCap
Aim #3 Adoption: Qualitative interviews | 12 weeks
  Semi-structured qualitative interviews will be conducted with patient, PT, support staff interviews regarding their lived experience integrating mindfulness and physical therapy. Analysis will generate qualitative themes that will be used to plan for a fully-powered trial.
Aim #3 Adoption: Mindfulness Oriented Recovery Enhancement component (MORE) | 12 weeks
  Percentage of patients enrolled after I-EPT training that report receiving any MORE component.
Aim #3 Implementation: Fidelity | 12 weeks
  Mindfulness Oriented Recovery Enhancement _functional measure (Modified MORE-FM) fidelity measure during patient encounters.
  The MORE FM will be completed by a rater which entails the reviewer listening to audio recordings of all patient encounters at the end of the 12 week patient management period.
  18-item scale - total scores range from 0 - 114. Scores are summed and averaged.
Aim #3 Implementation: Percentage of patients managed by PT | 12 weeks
  The percentage of patients managed by a single trained physical therapist (don't cross over between physical therapists)
Aim #3: Adoption, Maintenance and Implementation: Qualitative Interviews | 12 weeks
  Semi-structured qualitative interviews will be conducted with patient, PT, support staff, managers and clinic leadership interviews regarding their lived experience integrating mindfulness and physical therapy. These interviews will be used to understand potential barriers and facilitators for future adoption, implementation and maintenance of I-EPT
Aim #3: Physical therapist retention | 12 weeks
  The percentage of physical therapists who participate in the fidelity assessments
Aim #3: Patient retention | baseline, 6 weeks, 12 weeks
  Percentage of patients managed by study physical therapists who are retained at baseline, 6- and 12-week follow-up.
Aim #3: Screened patients | At recruitment
  Percentage of patients screened who are eligible
Sleep duration | baseline, 6 and 12 weeks
  hours and minutes of actual sleep during past month collected at baseline, 6 and 12 weeks
  We will also calculate the change from baseline to 6 weeks and the change from baseline to 12 weeks.
Aim # 3: Adoption: Patient retention | baseline, 6 and 12 weeks.
  Percentage of patients managed by study PTs who are retained at baseline, 6- and 12-week follow-up
Aim # 3 implementation: Modified version of the Mindfulness Oriented Recovery Enhancement - Functional Measure during patient encounters. | 12 weeks
  18 items. Scores range from 0 to 216. Higher scores equate to greater fidelity.
  Percentage of PTs who score an average of 3 on fidelity assessments
Aim #3: Adherence | 12 weeks
  THe number of recommended patient visits attended
Aim # 3 Adherence | weekly for 12 weeks
  Number of minutes spent practicing mindfulness, reappraisal or savoring each day
Aim # 3 Adoption: Patients receiving MORE Components | 12 weeks
  Percentage of patients enrolled that report receiving any MORE component

CONTACTS AND LOCATIONS:
Overall Officials: Jake Magel, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
1. The PI will provide data to outside researchers working under an institution with a federal wide assurance
  2. De-identified limited access data sets will be created and available for delivery through encrypted, password protected files
  3. To protect the confidentiality and privacy of the subjects, investigators granted access to these data must adhere to strict requirements. The Universities of Utah and Florida will define these requirements and establish criteria for access to data by outside researchers (as defined by current NIH regulations).
  4. We will make detailed versions of our standard operating procedures available to the scientific and clinical research community.
  5. Scientific publications will be the primary means of realeasing the analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 1 year after the completion of Aim 3
Access Criteria: The IDSA will be subject to review by both the University of Utah and University of Florida legal and IRB departments. Outside researchers will be required to submit approval from their own IRB. Conditions placed on the use of the data include
  1. No distribution to third parties
  2. Proper acknowledgment and citation of the data providers and grant funding
  3. Exclusive use by the data recipient in connection with a specific research project
  4. Data recipient will maintain ultimate responsibility for the data received
  5. Agreement not to use the data in any effort to establish the identity of participants
  6. Data recipient will be subject to applicable federal, state, and local laws or regulations and institutional policies providing additional protections for human subjects

REFERENCES:
- [Derived] Magel JS, Beneciuk JM, Siantz E, Fritz J, Garland EL, Hanley A, Shen J, Blosser P, Matev T, Gordon AJ. PT-IN-MIND: study protocol for a multisite randomised feasibility trial investigating physical therapy with integrated mindfulness (PT-IN-MIND) for patients with chronic musculoskeletal pain and long-term opioid treatment who attend outpatient physical therapy. BMJ Open. 2024 Jul 30;14(7):e082611. doi: 10.1136/bmjopen-2023-082611. PMID 39079926